CLINICAL TRIAL: NCT04274959
Title: Functional Evaluation of Ceramic Onlay Restorations With Different Preparation Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Mokhtar Nasr Sheded Alsedawy, lecturer assistant,fixed prosthodontics department,faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-02-01
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-09

CONDITIONS: Posterior Ceramic Onlays; Badly Decayed Teeth Need to be Restored , Teeth Restored With Large Filling Restorations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant, outcomes assessor) double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceramic onlay with shoulder preparation design. (Active Comparator): posterior ceramic onlay restoration with shoulder design with 1 mm shoulder thickness
  Interventions: Other: ceramic onlay with shoulder preparation design.
- ceramic onlay with butt joint preparation design (Experimental): posterior ceramic onlay with butt joint preparation design with flat occlusal reduction with inclined surface
  Interventions: Other: ,ceramic onlay with butt joint preparation design

INTERVENTIONS:
Other: ceramic onlay with shoulder preparation design. — ceramic onlay with shoulder preparation design which allowing the largest possible enamel for adhesion ,
  Arms: ceramic onlay with shoulder preparation design.
Other: ,ceramic onlay with butt joint preparation design — ceramic onlay with butt joint preparation design with cusp reduction to protect teeth from occlusal loads and cuspal fracture
  Arms: ceramic onlay with butt joint preparation design

SUMMARY:
Tooth preparation designs for posterior ceramic restorations have been based on traditional cast metal restoration designs, but with more occlusal tooth reduction and with a slightly increased taper. These preparations may involve the removal of considerable tooth structure. As more structure is removed, higher tooth strain and lower fracture resistance may occur.5 The increased tooth structure loss may increase cuspal flexure, thereby reducing the tooth fracture resistance, or open the restoration-tooth interface .

However, it has been demonstrated that cusp recovery results in fewer failures, likely increasing the longevity of posterior ceramic restorations. Recently, minimally invasive cavity preparations for posterior indirect restorations were demonstrated to present the benefit of conservation of tooth structure, as well as improved stress distribution. However, the performance of posterior restoration is also material dependent. Due to the continuous advancements in dental ceramics and innovative manufacturing techniques.

The aim of this study is to evaluate the clinical functional performance of ceramic onlay restorations with butt joint preparation design and compare them to shoulder preparation design.

DETAILED DESCRIPTION:
When an indirect restoration is selected as the treatment option for posterior teeth, the clinician must determine the configuration of the cavity preparation. Several designs have been proposed for preparing all-ceramic resin-bonded posterior restorations, as guided by the particular mechanical and structural characteristics of ceramic restorative materials. mechanical and structural characteristics of ceramic restorative materials. The primary causes of failure of ceramic onlay restorations are cohesive bulk fractures and marginal deficiencies, which manifest clinically as marginal discoloration and secondary caries. Tooth preparation designs for posterior ceramic restorations have been based on traditional cast metal restoration designs, but with more occlusal tooth reduction and with a slightly increased taper. These preparations may involve the removal of considerable tooth structure. As more structure is removed, higher tooth strain and lower fracture resistance may occur.5 The increased tooth structure loss may increase cuspal flexure, thereby reducing the tooth fracture resistance, or open the restoration-tooth interface .

However, it has been demonstrated that cusp recovery results in fewer failures, likely increasing the longevity of posterior ceramic restorations. Recently, minimally invasive cavity preparations for posterior indirect restorations were demonstrated to present the benefit of conservation of tooth structure, as well as improved stress distribution. However, the performance of posterior restoration is also material dependent. Due to the continuous advancements in dental ceramics and innovative manufacturing techniques.

Maximum preservation of sound tooth structure and maintenance of the vitality of restored teeth is critical for the longevity of teeth as well as restorations, especially in cases, where a large amount of tooth tissue has been lost due to wear and/or trauma. As the demand for conservative tooth treatment increases, so does the need for partial ceramic crowns. In addition to traditional cusp capping, simplified designs have been recommended in certain cases, such as fractured teeth and teeth with large caries.. According to the cusp coverage, the types of restorations can be classified as inlays, which is not covered cusps, onlays, which is covered at least one cusp, or overlays, and which is covered all cusps.

Onlay restorations not only provide superior esthetics but also minimize tooth tissue loss, making them a good treatment choice for posterior teeth with extensive cavities formed due to caries. Moreover, by covering more than one tooth cusp, onlays provide a favorable distribution of stress, reducing the risk of tooth and restoration fracture. preparation design may also play a role in tooth/restoration fracture. Some authors have shown that occlusal reduction reduces the chance of restoration failure. Others have shown that large preparation designs results in a reduced chance of possible fracture occurred in tooth tissue.

While different preparation designs have been described in the literature, the most appropriate design will vary according to the restorative material to be used. Despite the fact that partial ceramic crowns are increasingly advocated as alternative restorations for extensively damaged teeth, the literature includes limited studies examining the use of different preparation designs with this type of restoration. To date, confusing and contradictory results have been obtained regarding the effects of preparation design on the fracture resistance and stress distribution of tooth structure restored with partial ceramic crowns. Therefore, this study investigated the effects of three different preparation designs on the fracture of ceramic onlays. The hypothesis that different designs would affect the fracture resistance of onlay restorations.

ELIGIBILITY:
Inclusion Criteria:

* From 25-45 years old, be able to read and sign the informed consent document. (31)
* Have no active periodontal or pulpal diseases, have teeth with good restorations. (32)
* Psychologically and physically able to withstand conventional dental procedures
* Patients with teeth problems indicated for posterior onlay.

  1. Decayed teeth
  2. Teeth restored with large filling restorations
* Able to return for follow-up examinations and evaluation

Exclusion Criteria:

* Patient less than 25 or more than 45 years
* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene, high caries risk and uncooperative patients
* Pregnant women
* Patients in the growth stage with partially erupted teeth
* Psychiatric problems or unrealistic expectations
* Lack of opposing dentition in the area of interest.
* The presence of a removable or fixed orthodontic appliance, signs of bruxism or clenching, the absence of more than one unit in the posterior region .

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | 1 year
  measured using Modified united states public health service criteira (MUSPHS)

SECONDARY OUTCOMES:
Marginal adaptation | 1 year
  measured using Modified united states public health service criteira (MUSPHS)

OTHER OUTCOMES:
Patient satisfaction | 1year
  measured using(Questionnaire) VAS*(
  * Visual Analog Scale)

CONTACTS AND LOCATIONS:
Overall Officials: nora alsedawy, M.D.s, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No